CLINICAL TRIAL: NCT03530982
Title: Intensive Training of Functional Priorities Reported by Adolescents With Cerebral Palsy
Brief Title: Intensive Goal Training for Adolescents With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, MARINA B BRANDAO, Professor, Federal University of Minas Gerais
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 54597916.1.0000.5149
Record Dates: First submitted 2018-04-26; First posted 2018-05-21 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Individualized intensive training of functional priorities presented by adolescents with CP. The intervention will happen during 2 weeks, 5 days/week, during 3 hours in a local rehabilitation center. Trained occupational and physical therapists will conduct the intervention procedures
Masking Description: The assessor will not know the aims and content of the intervention procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Intensive goal training of relevant activities reported by adolescents in the beginning of the study. Therapists will grade the level of complexity of the proposed activities, considering the relevant movements, task demands and contextual factors involved in the performance of each task. Adolescents will be asked to practice these activities at home (1 hour/daily) and to discuss their difficulties and improvements with the therapists. The intervention will be provided in a day-camp model.
  Interventions: Other: Intensive goal training

INTERVENTIONS:
Other: Intensive goal training — Intensive goal training : 30 hours during 2 weeks
  Other Names: intensive individualized functional training

SUMMARY:
Adolescents with cerebral palsy (CP) present important limitations for the performance of daily living activities. The aims of the study is to evaluate the feasibility and effects of an intensive goal training protocol for adolescents with CP. He hypothesize that adolescents submitted to the studied protocol will present improvements in performance and satisfaction of prioritized functional goals.

DETAILED DESCRIPTION:
We will conduct a feasibility study to assess the implementation and the possible effects of an intensive individualized goal training with adolescents with CP. Adolescents will select up to 5 functional goals to be trained during a 2 weeks, 3 hour-daily training, totalling 30 hours across 2 weeks. Moreover, they will be asked to daily practice these activities at home along the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of bilateral CP;
* Age between 12 and 17 years old;
* Manual Ability Classification System (MACS) ranging from levels I to III;
* Gross Motor Function Classification System (GMFCS) ranging from levels I to IV;
* Ability to understand verbal instructions.

Exclusion Criteria:

* Botulinum toxin or surgery in upper limbs in the previous 6 months of the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2018-06-02 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Functional Goals | 1 month before intervention; pre-intervention; immediate post-intervention, 3-month follow-up
  Canadian Occupational Performance Measure (COPM) (ranging 1-10; higher values, better outcomes)
Change in Daily functioning- Self-Care | 1 month before intervention; pre-intervention; immediate post-intervention, 3-month follow-up
  Pediatric Evaluation Disability Inventory (PEDI) self-care: ranging from 0-63; higher values, better outcomes
Change in Daily functioning- Mobility | 1 month before intervention; pre-intervention; immediate post-intervention, 3-month follow-up
  Pediatric Evaluation Disability Inventory (PEDI) mobility: ranging from 0-55; higher values, better outcomes

SECONDARY OUTCOMES:
Change in Manual dexterity | 1 month before intervention; pre-intervention; immediate post-intervention, 3-month follow-up
  Box & Blocks Test (BBT)- number of blocks that are transported during 1 minute (there is no established max-min, higher values, better outcome)
Change in Gross motor function | 1 month before intervention; pre-intervention; immediate post-intervention, 3-month follow-up
  Gross Motor Function Measure (GMFM): gross motor function abilities assessed in activities from 5 domains: lying and rolling; seating; crawling and kneeling; standing; walking, running and jumping. higher scores, better outcome
Change in Participation at home | 1 month before intervention; pre-intervention; immediate post-intervention, 3-month follow-up
  Participation Environment Measure: Children and Youth (PEM-CY): Structured questionnaire to assess the frequency and level of involvement in daily living tasks (home scale will be used) higher scores, better outcomes
Change in Participation in household activities | 1 month before intervention; pre-intervention; immediate post-intervention, 3-month follow-up
  Children´s Helping Out: Responsibility, Expectations and Supports (CHORES): structured questionnaire to assess the frequency and level of assistance in household activities: higher scores, better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Associação Mineira de Reabilitação, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bleyenheuft Y, Ebner-Karestinos D, Surana B, Paradis J, Sidiropoulos A, Renders A, Friel KM, Brandao M, Rameckers E, Gordon AM. Intensive upper- and lower-extremity training for children with bilateral cerebral palsy: a quasi-randomized trial. Dev Med Child Neurol. 2017 Jun;59(6):625-633. doi: 10.1111/dmcn.13379. Epub 2017 Jan 30. PMID 28133725
- [Background] Charles J, Gordon AM. Development of hand-arm bimanual intensive training (HABIT) for improving bimanual coordination in children with hemiplegic cerebral palsy. Dev Med Child Neurol. 2006 Nov;48(11):931-6. doi: 10.1017/S0012162206002039. PMID 17044964
- [Background] de Brito Brandao M, Gordon AM, Mancini MC. Functional impact of constraint therapy and bimanual training in children with cerebral palsy: a randomized controlled trial. Am J Occup Ther. 2012 Nov-Dec;66(6):672-81. doi: 10.5014/ajot.2012.004622. PMID 23106987